CLINICAL TRIAL: NCT07144410
Title: Balancing Analgesia and Side Effects: Intrathecal Fentanyl and Morphine Versus Fentanyl for Cesarean Section Anesthesia
Brief Title: Pain Control and Side Effects in Cesarean Section Anesthesia: Comparison of Intrathecal Morphine and Fentanyl
Acronym: FvMinSACS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oradea (Other)
Collaborators: Oradea Pelican Clinic Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 08FvM_Medical Study
Record Dates: First submitted 2025-08-14; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anaesthesia, Spinal
Keywords: spinal anaesthesia; elective caesarean section; intrathecal opioids; fentanyl; morphine; opioids side effects; analgesia; fentanyl and morphine
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Morphine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fentanyl, Morphine and Bupivacaine: Pregnant patients scheduled for C-section that received a spinal anaesthesia mixture of Fentanyl, Morphine and Bupivacaine
  Interventions: Drug: fentanyl + morphine
- Fentanyl and Bupivacaine: Pregnant patients scheduled for C-section that received a spinal anaesthesia mixture of Fentanyl and Bupivacaine
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl + morphine — The purpose of the trial is to study the quality of anaesthesia and perioperative analgesia provided by fentanyl, morphine and bupivacaine versus fentanyl and bupivacaine, as well as their side effects.
  Other Names: plus bupivacaine
  Groups: Fentanyl, Morphine and Bupivacaine
Drug: fentanyl — The purpose of the trial is to study the quality of anaesthesia and perioperative analgesia provided by fentanyl, morphine and bupivacaine versus fentanyl and bupivacaine, as well as their side effects.
  Other Names: plus bupivacaine
  Groups: Fentanyl and Bupivacaine

SUMMARY:
Intrathecal opioids are frequently combined with local anesthetics to optimize spinal anesthesia for cesarean delivery. Fentanyl, a lipophilic opioid, offers rapid onset and enhanced intraoperative analgesia. However, its postoperative analgesic duration is limited, but in contrast, morphine, a hydrophilic opioid, provides prolonged postoperative pain control but has a slower onset and a higher incidence of adverse effects, notably nausea and vomiting. This prospective, randomized, double-blind, parallel study enrolled 180 parturients scheduled for elective cesarean section, all receiving spinal anesthesia with hyperbaric bupivacaine (7.5-10 mg, adjusted to height) plus either intrathecal fentanyl 25 µg (F group) or intrathecal morphine 100 µg and fentanyl 25µg (M+F group). Primary outcomes include intraoperative and postoperative pain scores, systemic opioid consumption, and patient satisfaction, while secondary outcomes assess the incidence of opioid-related side effects.

DETAILED DESCRIPTION:
Eligible patients will be allocated in a 1:1 ratio into one of two groups:

Group F (Fentanyl): Hyperbaric bupivacaine 0.5% combined with fentanyl 25 µg. Group M+F (Morphine + Fentanyl): Hyperbaric bupivacaine 0.5% combined with morphine 100 µg and fentanyl 25 µg.

The dose of hyperbaric bupivacaine (7.5-11 mg) will be determined according to patient height. Randomization will be performed using the envelope technique. Two anesthetists will participate in each case: The first anesthetist will perform the spinal anesthesia and will remain blinded to the drug solution. The second anesthetist will open the allocation envelope, prepare the assigned intrathecal solution, and provide it to the first anesthetist. All drugs will be sourced from the same manufacturer to ensure uniformity.

During the pre-anesthetic visit, all patients will receive detailed information regarding the aims of the study, the planned anesthetic technique, the postoperative analgesia regimen, and the use of the Numeric Pain Rating Scale (NPS). Demographic and clinical data will be collected, including height, term weight, age, smoking status, obstetric history (gesta/para), presence of preoperative contractions, full medical history, current medications, and any allergies.

An 18G intravenous cannula will be inserted, and 500 mL of Ringer lactate will be infused prior to anesthesia. All participants will fast preoperatively and will receive pantoprazole 40 mg and metoclopramide 10 mg as premedication.

Spinal anesthesia will be performed under aseptic conditions with the patient in the sitting position at the L3-L4 interspace using a 27G Whitacre needle via a midline approach. Local infiltration with 2 mL of 1% lidocaine will precede dural puncture. The anesthetic mixture will be injected manually at a rate of 1 mL per 15 seconds with a barbotage technique.

Following injection, patients will be placed in the supine position with left uterine displacement using a roll wedge under the right hip. Warmed Ringer lactate will be administered at a rate of 10-20 mL/kg/h throughout the perioperative period. All patients will wear anti-embolic stockings on the lower limbs.

Surgery will begin once sensory block (assessed by the cold test) reaches the T4 dermatome. Non-invasive blood pressure (BP) will be measured every minute until delivery and every 3-5 minutes thereafter; heart rate (HR) and oxygen saturation (SpO₂) will be continuously monitored. A systolic BP decrease below baseline will be treated with intravenous ephedrine 5-15 mg, repeated every minute as required until BP is restored. Oxytocin 5 IU will be administered intravenously at delivery, followed by additional doses if clinically indicated. Granisetron 1 mg IV and dexamethasone 4 mg IV will be administered at the start of surgery; granisetron 1 mg will be repeated 12 hours later. Additional antiemetics will be given as required.

Postoperative analgesia will be obtained by 1 g of Paracetamol every 6 hours and Ibuprofen 400 mg every 8 hours, administered either intravenously or orally. As a reserve pain control for high intesity pain Tramadol 50-100 mg IV will be given every 6 hours as required, with a maximum daily dose of 400 mg.

Data will be recorded for the following parameters:Demographic variables as age, weight, height, smoking status, obstetric history, preoperative contractions. Time from anesthesia induction to surgical incision, time to achieve sensory block.

Pain scores will be assessed at surgical incision, at the end of surgery, and postoperatively at 4, 6, 12, 24, 48, and 72 hours, both at rest and during mobilization. Side effects such as the incidence and severity of pruritus (graded), nausea, vomiting, oversedation, dizziness, and respiratory depression. Maximum motor block using the 4-point Bromage scale, time to complete motor recovery, and sensory block level determined by the cold test.

Pain intensity will be evaluated using the Numeric Pain Rating Scale (0 = no pain; 10 = worst pain imaginable) at all scheduled postoperative time points. But for a more comprehensively comparison of the post-operative pain in the study groups, two additional assessment metrics will be employed:

1. time-weighted sum pain intensity differences over 72 hours
2. sum pain intensity differences area over 72 hours Descriptive statistics will include the observed frequency counts (percentage) for categorical variables; and mean ± standard deviation for numerical variables, irrespective of their distribution. Normality will be tested with the Kolmogorov-Smirnov test. For comparing means in normally distributed values, the t-test for independent samples will be applied, with Levene's test for equality of variances. For comparing distribution of non-normally distributed numerical values, the non-parametric Mann-Whitney U statistical tests will be applied and median (Inter-Quartile Range) with Tukey's hinges will be additionally provided as a descriptive statistic.

The Chi-square statistical test (either asymptotic, Fisher's exact test, or Monte-Carlo simulation with 10,000 samples) will be applied to check the statistical significance of the association between the categorical variables. The odds ratio (OR) values will be calculated for the symptoms associated with the two anesthetics, such as nausea and dizziness.

The statistical analysis will be conducted at a 95% level of confidence and a 5% level of statistical significance. All reported probability values will be two-tailed.

Statistical analysis will be performed with the statistical software IBM SPSS v. 20 and open source R v.4.0.5 packages.The study will be conducted in accordance with the Declaration of Helsinki, and the protocol was approved by the Ethics Committees of Pelican Hospital from Oradea (no.1689/25.08.2025).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class I-II.
* Absence of significant past medical conditions.
* No documented hypersensitivity to any study drug.
* No history of chronic pain syndromes or regular analgesic consumption.
* No anxiety or depressive disorders diagnosis.
* Body weight ≥ 50 kg.
* Scheduled for elective cesarean delivery.
* Single fetus.

Exclusion Criteria:

* Patient refusal.
* Contraindication of spinal anaesthesia.
* Conversion from a natural delivery with or without an epidural anaesthesia started.
* History of substance abuse or drug dependence.
* Presence of acute or chronic fetal distress.
* Preeclampsia.
* Allergic reaction occurring after enrollment.
* Refusal to receive protocol-specified analgesics or medications.
* Requirement for surgical re-intervention within 72 hours postoperatively.
* Previous administration of opioids or other central nervous system depressants prior to intervention.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: The subjects of the study will be selected from the pregnant patients of Oradea Pelican Clinic Hospital.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Assessing the perioperative analgesic efficacy | 6 months
  Pain intensity will be evaluated using the Numeric Pain Scale, with scores obtained at the time of skin incision, at the end of surgery, and at 4h, 6h, 12h, 24h, 48h, and 72 hours postoperatively; AUE72h (sum pain intensity differences area over 72 hours) and SPID72h (time-weighted sum pain intensity differences over 72 hours). Assessments will be conducted both at rest and during mobilization. The pain scores according to the Numeric Pain Scale will be rated between 0 and 10, meaning 0 - no pain and 10 - the worst pain imaginable
Assessing the degree of patient's satisfaction | 6 months
  Assessing the degree of satisfaction on a five point scale with the highest rate as being "completely satisfied", followed by "satisfied", "so so", "unsatisfied" and "completely unsatisfied"

SECONDARY OUTCOMES:
Incidence of Additional Opioid-Related Adverse Effects | 6 months
  Other potential opioid-related adverse effects, including nausea, vomiting, dizziness, sedation, and respiratory depression, will be documented as present or absent during the first 72 postoperative hours.
Incidence and Severity of Pruritus | 6 months
  Pruritus associated with intrathecal opioid administration will be recorded and graded on a 4-point scale: 0 - absent; 1 - mild; 2 - moderate; 3 - severe.

CONTACTS AND LOCATIONS:
Overall Officials: Aurel Mohan, MD, PhD, Study Chair — Head of Surgery Department of Medicine and Pharmacy Faculty of Oradea
Locations (1):
- University of Oradea, Pelican Clinic Hospital, Oradea, Bihor County, Romania